CLINICAL TRIAL: NCT00391326
Title: Efficacy and Safety of Prehospital Administration of Bivalirudin in STEMI Patients Redirected for Primary PCI Based on Tele-Transmitted 12-Lead ECGs
Brief Title: Efficacy and Safety of Prehospital Administration of Bivalirudin in STEMI Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: H:S Laegeambulance (Other)
Responsible Party: Peter Clemmensen, Rigshospitalet
Other Study IDs: J.nr. 2006-41-6849
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Bivalirudin; Heparin; Bleeding; TIMI flow; STEMI
MeSH Terms: conditions — Hemorrhage; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the efficacy and safety of prehospital administration of bivalirudin, as a substitute for heparin, in patients with acute myocardial infarction redirected for primary angioplasty bypassing local hospitals, immediately after the diagnosis is confirmed via tele-transmission of a 12-lead electrocardiogram.

DETAILED DESCRIPTION:
Primary angioplasty (pPCI) is the therapy of choice in patients with ST elevation acute myocardial infarction (STEMI) in Denmark. However, time is lost transferring patients from a local hospital to an invasive treatment centre. Time can be saved by redirecting STEMI patients to pPCI based on wireless prehospital 12-lead electrocardiogram (ECG) transmission directly to a cardiologist's handheld device. To prevent complications during the transportation of STEMI patients to the invasive hospital, patients are treated with oxygen, aspirin, clopidogrel, heparin, and nitro-glycerine in the ambulance. However, heparin use is cumbersome for the ambulance personnel since it must be kept at 5 degrees Celsius. An alternative to heparin may be bivalirudin, since it can be kept at room temperature and thus is easily administered in the prehospital setting.

Comparison: Heparin versus bivalirudin treatment. Efficacy is determined by thrombolysis in myocardial infarction (TIMI) flow in the first and final coronary angiogram. Safety is determined by the rate of bleeding complication.

ELIGIBILITY:
Inclusion Criteria:

* ST elevation acute myocardial infarction patients redirected for primary angioplasty
* Symptoms less than 12 hours

Exclusion Criteria:

* Contraindications against primary angioplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with STEMI transferred directly to primary PCI based og transmission of a prehospital ECG
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Clemmsensen, MD. phD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - H:S Lægeambulance, Copenhagen, V
  - Rigshospitalet, Copenhagen, Ø